CLINICAL TRIAL: NCT06517784
Title: Insulin Initiation and Adherence Behaviours: a Cross Sectional Survey of Indian HCPs & Patients With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN000-7941; U1111-1302-7518 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-07-18; First posted 2024-07-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with type 2 diabetes
  Interventions: Other: No treatment given
- Health care providers: Health care providers who treat patients with type 2 diabetes
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
This is a cross-sectional study planned among patients with Type 2 Diabetes (T2D) and Health Care Providers (HCPs) who treat T2D patients. Study participants will be recruited through existing databases/panels to complete a 30-minute self-administered online survey. The purpose of the study is to understand the insulinization barriers and the insulin adherence behaviours of both HCPs and patients.

ELIGIBILITY:
Inclusion Criteria:

For patients

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Diagnosed with T2D
4. Currently seeing an HCP for T2D
5. Initiated on insulin within the past 12 months
6. Prescribed insulin on a permanent basis
7. Currently taking insulin via a vial and syringe or insulin pen

For HCP

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Primary care physician (PCP) with degree in internal medicine or general medicine, diabetologist with degree in internal medicine or general medicine plus diploma in diabetology, or endocrinologist
4. Has been in practice a minimum of 2 years
5. Diabetologist/endocrinologist: treats at least 50 T2D patients per month
6. PCP: treats at least 40 T2D patients per month
7. Currently initiates T2D patients on insulin
8. Treats 20 percent or more of T2D patients with insulin

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes (T2D) and Health Care Providers (HCPs) who treat T2D patients
Sampling Method: Non-Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
The barriers toward insulin initiation among HCPs & patients | At time of data abstraction (Day 1)
  Barriers to insulin initiation = Likert scale: 1=Strongly disagree, 5=Strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk India, Bangalore, India

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com